CLINICAL TRIAL: NCT00538330
Title: Post Operative Adjuvant Chemotherapy Followed by Adjuvant Tamoxifen vs Nil for Patients With Operable Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RAC #93-107
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen

SUMMARY:
Post operative adjuvant chemotherapy followed by adjuvant Tamoxifen vs nil for patients with operable breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with operable breast cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2007-09; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
safety | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Ezzat, MD, Principal Investigator — KFSH&RC, Riyadh